CLINICAL TRIAL: NCT05513911
Title: Intermittent Hypoxia and Upper Limb Training in Individuals With Spinal Cord Injury
Brief Title: Intermittent Hypoxia and Upper Extremity EMG Recordings in Individuals With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00201602
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries
Keywords: Acute Intermittent Hypoxia; Motor Unit; Upper Extremity
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Insemination, Artificial, Homologous

STUDY DESIGN:
Intervention Model Description: Every participant in this study will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute intermittent Hypoxia Therapy (Experimental): This group will receive the acute intermittent hypoxia therapy (9% O2) for 30 minutes. Before and after the intervention the participant will perform flexion of the elbow at various levels of intensity
  Interventions: Other: Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — Acute Intermittent Hypoxia is administered in 30-60 second bouts of 9% O2 concentration, followed by 60-90 seconds of normoxic air concentrations (21% O2, room air). This procedure is repeated 15 times for a 30 minute session
  Other Names: AIH

SUMMARY:
In this current study, the examiners examine some of the mechanisms of how Acute Intermittent Hypoxia (AIH) effects the upper extremity of survivors of spinal cord injury. This is accomplished both with the use of a load cell to determine elbow strength changes and high density grid electromyography (EMG) to record bicep muscle activations before and after bouts of AIH

DETAILED DESCRIPTION:
It has been shown previously that there is an increase in strength in survivors of spinal cord injury after brief bouts of Acute Intermittent Hypoxia. In this study, participants are fitted with a high density EMG electrode on the biceps brachii, and attached to a load cell at the wrist, they are asked to flex and extend their elbow at various levels of intensity. This is performed before and after the 30 minute session of AIH. The investigators hope to identify specific types of motor units of the upper extremity of survivors of spinal cord injury after AIH to help further our understanding of what mechanisms may be causing the known increase in muscle strength post AIH

ELIGIBILITY:
Inclusion Criteria:

* History of Spinal Cord Injury from C3-T4
* Non-progressive spinal cord injury
* More than 6 months since initial Spinal Cord injury
* Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

* Presence of any of the following medical conditions: Congestive heart failure, arrhythmia, uncontrolled high blood pressure, uncontrolled diabetes mellitus, COPD/emphysema and severe asthma
* Persons with known coronary artery disease, a history of myocardial infarction, or known carotid or intracerebral artery stenosis
* Medical clearance will be required if participant is taking any other investigational agents
* Women who are pregnant or nursing
* Individuals with tracheostomy
* Cannot pursue other research studies which may interfere
* Unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Maximal Elbow Strength [Newtons] | 30 minutes Post intervention
  Recordings of the elbow joint torque are taken while the participant is asked to flex and extend the elbow voluntarily at a maximum level of intensity

SECONDARY OUTCOMES:
Biceps Brachii Muscle activation [μv] | 30 minutes post intervention
  Peak electromyographic activation of the biceps brachii muscle during maximum voluntary flexion and extension tasks

CONTACTS AND LOCATIONS:
Overall Officials: William Z Rymer, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab; Milap Sandhu, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Overall participant Data will be reported in publications